CLINICAL TRIAL: NCT06478134
Title: Efficacy and Safety of a Multiple-Action Tear Substitute (TriMix) in Dry Eye Disease: A Randomized, Double-blinded, HA-controlled Study
Brief Title: Efficacy and Safety of a Multiple-Action Tear Substitute (TriMix) in Dry Eye Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, José-María Sánchez-González, OD, PhD, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIVIUS-ABS-002
Record Dates: First submitted 2024-06-14; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Patients were instructed to instill 1 drop TriMix tear substitute or 0.15% HA tear substitute into each eye 3 times per day for 6 months. HA-based tear substitutes can reduce tear film hyperosmolarity and are effective in treating DED. Therefore, 0.15% HA tear substitute was selected as a suitable comparator.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: TriMix tear substitute and 0.15% HA tear substitute are transparent, with no special smell and the bottles were identical in appearance such that patients, investigators and care provider were masked to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TriMix (Experimental): A new-generation tear substitute containing cross-linked hyaluronic acid 0.15%, trehalose 3%, liposomes 1% and sterylamine 0.25%.
  Interventions: Drug: Trimix tear substitutes
- Hyaluronic acid (Active Comparator): 0.15% Hyaluronic acid tear substitute.
  Interventions: Drug: Hyaluronic acid tear substitute

INTERVENTIONS:
Drug: Trimix tear substitutes — Patients were instructed to instill 1 drop of TriMix tear substitute into each eye 3 times per day for 6 months.
  Arms: TriMix
Drug: Hyaluronic acid tear substitute — Patients were instructed to instill 1 drop of 0.15% HA tear substitute into each eye 3 times per day for 6 months.
  Arms: Hyaluronic acid

SUMMARY:
The objective of the study is to assess the efficacy and safety of TriMix tear substitute in patients with dry eye disease. For this purpose, a randomized, double-blind clinical trial has been designed, using an Hyaluronic acid-based tear substitute as a control.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported history DED while working with computer screens ≥ 6 hours per day.
2. ocular surface disease index (OSDI) > 13 points.
3. non-invasive tear film break-up time (NIBUT) < 10 s.
4. Schirmer test (ST) without anesthesia ≥ 5 mm.
5. MGD grade ≤ 1. For MGD, the Sirius device (CSO, Florence, Italy) was used, which determines MGD grade based on loss area of meibomian glands (LAMG). MGD grade was scored from 0 to 4 (MGD grade 1 = LAMG < 25%; MGD grade 2 = LAMG ≥ 25% and < 50%; MGD grade 3 = LAMG ≥ 50% and < 75%; MGD grade 4 = LAMG ≥ 75%).

Exclusion Criteria:

1. abnormal lid anatomy, including active blepharitis, and active lid margin.
2. all corneal disorders that affect diagnostic test, such as active corneal infection and corneal dystrophies.
3. active ocular allergies.
4. vectored thermal pulsation (VTP) intense pulse light (IPL), quantum molecular resonance (QMR), or other procedure to treat DED within the previous 6 months.
5. intraocular surgery or laser ocular surgery within the previous 6 months.
6. use of topical antibiotics and anti-inflammatory treatments, including steroids and non-steroidal anti-inflammatory drugs.
7. systemic autoimmune diseases.
8. contact lens wearers.
9. pregnant or lactating women.
10. patients who did not understand or comprehend the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Ocular surface disease index questionnaire | This outcome measure was analyzed at baseline, 3 months and 6 months.
  The OSDI questionnaire were employed to assess the severity of DED symptoms, with scores ranging from 0 (indicating no ocular surface disease) to 100 (indicating severe ocular surface disease) points. This questionnaire was provided during consultations at each follow-up visit.
Non-invasive tear film break-up time | This outcome measure was analyzed at baseline, 3 months and 6 months.
  Tear film stability was automatically assessed using NIBUT by projecting Placido rings from the Sirius device (CSO, Florence, Italy) onto the corneal surface. The time interval between the last blink and the initial distortion of the ring pattern was defined as first NIBUT. This variable was always measured at least 12 hours after administration of the study medication and the average of 3 consecutive measurements was calculated for statistical analysis.
Schirmer I test without anesthesia | This outcome measure was analyzed at baseline, 3 months and 6 months.
  During the test, the patient is instructed to look upward while the test strip is carefully positioned between the palpebral conjunctiva of the lower eyelid and the bulbar conjunctiva. Subsequently, the patient is asked to keep their eyes gently closed for five minutes. After this period, the test strip is removed, and the Schirmer test score is determined by measuring the length of the moistened area on the strip.

CONTACTS AND LOCATIONS:
Overall Officials: José-María Sánchez-González, Study Director — University of Seville
Locations (1):
- Novovision ophthalmologic clinic, Murcia, Spain

REFERENCES:
- [Background] Vigo L, Senni C, Pellegrini M, Vagge A, Ferro Desideri L, Carones F, Scorcia V, Giannaccare G. Effects of a New Formulation of Multiple-Action Tear Substitute on Objective Ocular Surface Parameters and Ocular Discomfort Symptoms in Patients with Dry Eye Disease. Ophthalmol Ther. 2022 Aug;11(4):1441-1447. doi: 10.1007/s40123-022-00518-7. Epub 2022 May 14. PMID 35567735
- [Background] Roszkowska AM, Inferrera L, Spinella R, Postorino EI, Gargano R, Oliverio GW, Aragona P. Clinical Efficacy, Tolerability and Safety of a New Multiple-Action Eyedrop in Subjects with Moderate to Severe Dry Eye. J Clin Med. 2022 Nov 26;11(23):6975. doi: 10.3390/jcm11236975. PMID 36498550

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT06478134/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT06478134/ICF_001.pdf